CLINICAL TRIAL: NCT04064866
Title: A Multi-Center, Randomized, Controlled, Double-blind Study Evaluating Safety and Efficacy of Hemocyte Autograft for Treatment of Single-Level and Multi- Level Lumbar, Thoracic and Cervical Discogenic Pain
Brief Title: Safety and Efficacy of PRP for Treatment of Disc Pain
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Neurological Associates of West Los Angeles (Other)
Collaborators: EmCyte Corporation (Industry); BioRich Medical (Unknown)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Quadruple | Purpose: Treatment
Other Study IDs: 31135/1
Record Dates: First submitted 2019-08-19; First posted 2019-08-22 (Actual); Last update posted 2019-12-04 (Actual); Status verified 2019-12

CONDITIONS: Discogenic Pain
Keywords: Lumbar Spine; Thoracic Spine; Cervical Spine

STUDY DESIGN:
Intervention Model Description: This is a multi-center, randomized, controlled, double-blind clinical trial comparing hemocyte autograft (platelet rich plasma) to control injection (placebo) in subjects with reported cervical, thoracic or lumbar pain for at least 3 months with Pfirrmann grade changes at 7 or less and who are being considered for discography in order to identify pain generator discs in evaluation of potential surgical candidates. Randomization ratio was 2:1. After 8 weeks subjects who received placebo are eligible for crossover to treatment arm with hemocyte autograft, and subject who received treatment arm are eligible for surgery if not improved.
  For subjects who cross over, follow-up schedule will reset with visits at 8 weeks and 26 weeks post-crossover.
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Masking Description: Investigator, care provider, and participant were all blinded to injection contents (e.g., hemocyte autograft intervention vs. placebo control) An independent blinded evaluator assessed subjects at 4 weeks and 8 weeks. An unblinded or blinded evaluator will assess subjects at 26 weeks.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: Yes

ARMS (2):
- PRP/Hemocyte Autograft Intervention Arm (Experimental): All subjects will have blood drawn (50 cc) from any access site and have it prepared for hemocyte autograft. Using a 20 gauge introducer and 25 gauge disc needle, subjects randomized to active condition will have exactly 3 cc of hemocyte autograft placed in a 3 cc syringe. The syringe barrels and tubing were covered with opaque tape so that the injector was blinded to the contents. 1-2 cc of PRP was injected into the nucleus pulposus of each identified treatment level disc for lumbar; 0.5-1 cc for thoracic and 0.5-1 cc for cervical.
  Interventions: Device: High yield pure PRP; Device: ProPlaz PPC
- Placebo Control Arm (Placebo Comparator): All subjects will have blood drawn (50 cc) from any access site and have it prepared for hemocyte autograft. Using a 20 gauge introducer and 25 gauge disc needle, subjects randomized to placebo condition will have exactly 3 cc of saline placed in a 3 cc syringe. 1-2 cc of saline was injected into the nucleus pulposus of each identified treatment level disc for lumbar; 0.5-1 cc for thoracic and 0.5-1 cc for cervical.
  Interventions: Other: Placebo

INTERVENTIONS:
Device: High yield pure PRP — The investigational product is hemocyte autograft derived from the subject's own blood. Subjects with a clinical diagnosis of discogenic pain had a discogram with ¼ cc to ½ cc of contrast injected by hand (leaving up to ½ cc contrast in the needle lumen and connecting tube); any concordant pain will be noted. Subjects received the injectant delineated by coordinator-provided randomization. Subjects were awake for the entirety of study treatment procedure.
  All subjects had blood drawn (50 cc) from any access site and double-centrifuged using the EmCyte Hemocyte Autograft system; the first spin separated the buffy coat, the second spin and subsequent siphoning separated a purified platelet sample.
  Other Names: PRP
  Arms: PRP/Hemocyte Autograft Intervention Arm
Other: Placebo — Placebo injections will have saline placed in centrifuges and run for the duration required for PRP preparation. 3cc of saline will be placed in 3 cc syringes with opaque tape around the barrel to cover the fluid chamber. 1-2 cc of saline will be injected into the nucleus pulposus of each treatment level disc under fluoroscopy for lumbar; 0.5-1 cc for thoracic and 0.5-1 cc for cervical.
  Other Names: Control
  Arms: Placebo Control Arm
Device: ProPlaz PPC — Trademarked name of an FDA-cleared product
  Other Names: BioRich Medical ProPlaz Protein Plasma Concentrator
  Arms: PRP/Hemocyte Autograft Intervention Arm

SUMMARY:
This is a multi-center, randomized, controlled, double-blind clinical trial comparing hemocyte autograft (platelet rich plasma) to control injection (placebo) in subjects with reported cervical, thoracic or lumbar pain for at least 3 months with Pfirrmann grade changes at 7 or less and who are being considered for discography in order to identify pain generator discs in evaluation of potential surgical candidates.

DETAILED DESCRIPTION:
The study will recruit 180 subjects: 60 suffering from lumbar discogenic pain, 60 suffering from thoracic discogenic pain and 60 suffering from cervical discogenic pain. In each arm 40 study subjects will be randomized to receive hemocyte autograft, while 20 will be randomized to receive contrast as the control group. All subjects will have blood drawn (50 cc) from any access site and have it prepared for hemocyte autograft. Using a 20 gauge introducer and 25 gauge disc needle, subjects randomized to active condition will have exactly 3 cc of hemocyte autograft placed in a 3 cc syringe while subjects randomized to placebo will have exactly 3 cc of saline placed in a 3 cc syringe. The syringe barrels and tubing will be completely covered with opaque tape so that the injector is blinded to the contents. For both conditions, 1-2 cc of designated injectant (PRP for active, saline for placebo) will be injected into the nucleus pulposus of each identified treatment level disc for lumbar; 0.5-1 cc for thoracic and 0.5-1 cc for cervical. Primary endpoint will be at 8 weeks after injection. After 8 weeks subjects who received placebo are eligible for crossover to treatment arm with hemocyte autograft, and subject who received treatment arm are eligible for surgery if not improved.

ELIGIBILITY:
Inclusion Criteria:

1. Male or Female at least 18 years of age.
2. Clinically suspected discogenic pain in the cervical, thoracic or lumbar spine.
3. Bring considered for discography in order to identify source of pain in the evaluation of potential surgical candidates.
4. History of neck pain or mid or low back pain for at least 3 months.
5. Failed to respond to conservative therapies that include physical therapy and analgesics.
6. Documented Pfirrmann grade changes of 7 or less at each treatment level as represented by an MRI no more than 12 months old (extravasation not excluded).

Exclusion Criteria:

1. Unresolved neck or back pain from a previous cervical, thoracic or lumbar surgery at any level.
2. Any contraindication for discography or surgery
3. Significant signs or symptoms of root or cord compression at treatment levels.
4. Any diagnosis of a concurrent pain disorder or other concurrent cause of disability.
5. Daily opioid requirements of greater than180 mg oral morphine equivalent

   (OME) per day.
6. Current active systemic infection, or history of disc infection.
7. Untreated disabling thought or mood disorder.
8. Inability to provide informed consent including subjects in a socially compromised condition such as prisoners.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 27 (Actual)
Dates: Start 2016-05-17 (Actual); Primary Completion 2018-12-31 (Actual); Study Completion 2019-02-18 (Actual)

PRIMARY OUTCOMES:
Patient Specific Functional Scale (PSFS) | 8 weeks from baseline
  The primary objective of this study is to determine safety and efficacy of a single injection of hemocyte autograft into diseased discs for the treatment of back and neck pain. The PSFS is a self-report, patient-specific outcome measure designed to assess functional change in patients with pain and musculoskeletal disorders. The total score = the sum of the activity scores (10 maximum, which reflects a better level of functioning)/the number of activities (7 maximum). At least two points improvement on the average Pain Specific Functional
  Scale (PSFS).
Adverse Event Reporting | Baseline to 26 weeks
  Adverse events (AEs) and any other untoward signs or symptoms were collected at each study timepoint starting at the treatment injection. Serious adverse events (SAEs) determined by the investigator to be related to the study treatment were formally recorded. [NOTE: NONE REPORTED THROUGHOUT STUDY DURATION]

SECONDARY OUTCOMES:
Numeric Pain Rating Scale (NRPS) | 8 weeks from baseline
  The NRPS is a unidimensional measure of pain intensity for adults. The 11-point numeric scale ranges from '0' representing 'no pain' to 10 representing 'worst possible pain.' The NPRS can be administered verbally or graphically for self-completion. The respondent is asked to indicate the numeric scale value that best describes the intensity of their pain within the last 24-hours. Clinical improvement was denoted by at least 3 points improvement in Numeric Pain Rating Scale (NPRS)
Oswestry Disability Index (ODI) | 8 weeks from baseline
  A measure to gauge improvement in pain symptoms among lumbar and thoracic spine conditions. The ODI is a patient-based questionnaire which gives a subjective percentage score of functionality/disability for a list of activities of daily living among those rehabilitating from lower back pain. There are 6 statements scored from 0-5 (0 is the least pain/no pain, 5 is the greatest level of pain). Clinical improvement is characterized by more than 10% improvement in the ODI from baseline (calculated by [total scored/total possible score]*100).
Neck Disability Index (NDI) | 8 weeks from baseline
  The most commonly-used self-report measure to gauge improvement in pain symptoms among cervical spine conditions. The NDI is comprised of 10 items (each scored on a 0-5 rating scale, in which zero reflects "no pain" and five means "worst pain imaginable") including pain, personal care, reading, lifting, headaches, concentration, work ,driving, sleeping, and recreation. A higher score indicates greater level of disability. The NDI can be scored as a raw score of doubled and expressed as a percentile. 0-4 points (0-8%) = no disability. 5-14 points (10-28%) = mild disability. 15-24 points (30-48%) = moderate disability. 25-34 points (50-64%) = severe disability. 35-50 point (70-100%) = complete disability. Clinical improvement was indicated by improvement of at least 10% from baseline.

CONTACTS AND LOCATIONS:
Overall Officials: Sheldon E Jordan, M.D., Principal Investigator — Neurological Associates of West Los Angeles
Locations (7):
- United States (7):
  - Comprehensive Spine and Sports Center, Campbell, California
  - Neurological Associates of West LA, Santa Monica, California
  - The Spine Institute: Center for Spinal Restoration, Santa Monica, California
  - Thrive Treatment, Santa Monica, California
  - Georgia Pain and Spine, Peachtree City, Georgia
  - Millenium Pain Center, Chicago, Illinois
  - Precision Spine Care, Tyler, Texas

REFERENCES:
- [Background] Terry, A., Lutz, G., et al. Lumbar Intradiscal Platelet Rich Plasma Injections: A Prospective, Double-Blind, Randomized Controlled Trial. (2013), International Spine Intervention Society - 2013 21st Annual Scientific Meeting Research Abstracts. Pain Medicine, 14: 1269-1276. doi: 10.1111/pme.12219, 2013.
- [Background] Hoy D, March L, Brooks P, Blyth F, Woolf A, Bain C, Williams G, Smith E, Vos T, Barendregt J, Murray C, Burstein R, Buchbinder R. The global burden of low back pain: estimates from the Global Burden of Disease 2010 study. Ann Rheum Dis. 2014 Jun;73(6):968-74. doi: 10.1136/annrheumdis-2013-204428. Epub 2014 Mar 24. PMID 24665116
- [Background] Foster TE, Puskas BL, Mandelbaum BR, Gerhardt MB, Rodeo SA. Platelet-rich plasma: from basic science to clinical applications. Am J Sports Med. 2009 Nov;37(11):2259-72. doi: 10.1177/0363546509349921. PMID 19875361
- [Background] Pavlovic V, Ciric M, Jovanovic V, Stojanovic P. Platelet Rich Plasma: a short overview of certain bioactive components. Open Med (Wars). 2016 Aug 12;11(1):242-247. doi: 10.1515/med-2016-0048. eCollection 2016. PMID 28352802
- [Background] Boswell SG, Cole BJ, Sundman EA, Karas V, Fortier LA. Platelet-rich plasma: a milieu of bioactive factors. Arthroscopy. 2012 Mar;28(3):429-39. doi: 10.1016/j.arthro.2011.10.018. Epub 2012 Jan 28. PMID 22284405
- [Background] Blair P, Flaumenhaft R. Platelet alpha-granules: basic biology and clinical correlates. Blood Rev. 2009 Jul;23(4):177-89. doi: 10.1016/j.blre.2009.04.001. Epub 2009 May 17. PMID 19450911
- [Background] Sanchez AR, Sheridan PJ, Kupp LI. Is platelet-rich plasma the perfect enhancement factor? A current review. Int J Oral Maxillofac Implants. 2003 Jan-Feb;18(1):93-103. PMID 12608674
- [Background] Peng BG. Pathophysiology, diagnosis, and treatment of discogenic low back pain. World J Orthop. 2013 Apr 18;4(2):42-52. doi: 10.5312/wjo.v4.i2.42. Print 2013 Apr 18. PMID 23610750
- [Background] Wang SZ, Rui YF, Tan Q, Wang C. Enhancing intervertebral disc repair and regeneration through biology: platelet-rich plasma as an alternative strategy. Arthritis Res Ther. 2013;15(5):220. doi: 10.1186/ar4353. PMID 24165687
- [Background] Anitua E, Padilla S. Biologic therapies to enhance intervertebral disc repair. Regen Med. 2018 Jan;13(1):55-72. doi: 10.2217/rme-2017-0111. Epub 2018 Jan 22. PMID 29355455
- [Background] Davis VL, Abukabda AB, Radio NM, Witt-Enderby PA, Clafshenkel WP, Cairone JV, Rutkowski JL. Platelet-rich preparations to improve healing. Part I: workable options for every size practice. J Oral Implantol. 2014 Aug;40(4):500-10. doi: 10.1563/AAID-JOI-D-12-00104. PMID 25106016
- [Background] Li P, Zhang R, Zhou Q. Efficacy of Platelet-Rich Plasma in Retarding Intervertebral Disc Degeneration: A Meta-Analysis of Animal Studies. Biomed Res Int. 2017;2017:7919201. doi: 10.1155/2017/7919201. Epub 2017 Jul 2. PMID 28752097
- [Background] Gelalis ID, Christoforou G, Charchanti A, Gkiatas I, Pakos E, Papadopoulos D, Ploumis A, Korompilias A. Autologous platelet-rich plasma (PRP) effect on intervertebral disc restoration: an experimental rabbit model. Eur J Orthop Surg Traumatol. 2019 Apr;29(3):545-551. doi: 10.1007/s00590-018-2337-1. Epub 2018 Oct 28. PMID 30370433
- [Background] Khalaf K, Nikkhoo M, Ya-Wen Kuo, Yu-Chun Hsu, Parnianpour M, Campbell-Kyureghyan N, Haghpanahi M, Jaw-Lin Wang. Recovering the mechanical properties of denatured intervertebral discs through Platelet-Rich Plasma therapy. Annu Int Conf IEEE Eng Med Biol Soc. 2015 Aug;2015:933-6. doi: 10.1109/EMBC.2015.7318516. PMID 26736416
- [Background] Marx RE. Platelet-rich plasma: evidence to support its use. J Oral Maxillofac Surg. 2004 Apr;62(4):489-96. doi: 10.1016/j.joms.2003.12.003. No abstract available. PMID 15085519
- [Background] Tuakli-Wosornu YA, Terry A, Boachie-Adjei K, Harrison JR, Gribbin CK, LaSalle EE, Nguyen JT, Solomon JL, Lutz GE. Lumbar Intradiskal Platelet-Rich Plasma (PRP) Injections: A Prospective, Double-Blind, Randomized Controlled Study. PM R. 2016 Jan;8(1):1-10; quiz 10. doi: 10.1016/j.pmrj.2015.08.010. Epub 2015 Aug 24. PMID 26314234
- [Background] Fujita N, Imai J, Suzuki T, Yamada M, Ninomiya K, Miyamoto K, Iwasaki R, Morioka H, Matsumoto M, Chiba K, Watanabe S, Suda T, Toyama Y, Miyamoto T. Vascular endothelial growth factor-A is a survival factor for nucleus pulposus cells in the intervertebral disc. Biochem Biophys Res Commun. 2008 Jul 25;372(2):367-72. doi: 10.1016/j.bbrc.2008.05.044. Epub 2008 May 19. PMID 18492486
- [Background] Yazawa M, Ogata H, Nakajima T, Mori T, Watanabe N, Handa M. Basic studies on the clinical applications of platelet-rich plasma. Cell Transplant. 2003;12(5):509-18. doi: 10.3727/000000003108747073. PMID 12953925
- [Background] Everts PA, Malanga GA, Paul RV, Rothenberg JB, Stephens N, Mautner KR. Assessing clinical implications and perspectives of the pathophysiological effects of erythrocytes and plasma free hemoglobin in autologous biologics for use in musculoskeletal regenerative medicine therapies. A review. Regen Ther. 2019 May 10;11:56-64. doi: 10.1016/j.reth.2019.03.009. eCollection 2019 Dec. PMID 31193111
- [Background] Hussain N, Johal H, Bhandari M. An evidence-based evaluation on the use of platelet rich plasma in orthopedics - a review of the literature. SICOT J. 2017;3:57. doi: 10.1051/sicotj/2017036. Epub 2017 Oct 9. PMID 28990574
- [Background] Sanapati J, Manchikanti L, Atluri S, Jordan S, Albers SL, Pappolla MA, Kaye AD, Candido KD, Pampati V, Hirsch JA. Do Regenerative Medicine Therapies Provide Long-Term Relief in Chronic Low Back Pain: A Systematic Review and Metaanalysis. Pain Physician. 2018 Nov;21(6):515-540. PMID 30508983
- [Background] van Hooff ML, Spruit M, Fairbank JC, van Limbeek J, Jacobs WC. The Oswestry Disability Index (version 2.1a): validation of a Dutch language version. Spine (Phila Pa 1976). 2015 Jan 15;40(2):E83-90. doi: 10.1097/BRS.0000000000000683. PMID 25575092
- [Background] Childs JD, Piva SR, Fritz JM. Responsiveness of the numeric pain rating scale in patients with low back pain. Spine (Phila Pa 1976). 2005 Jun 1;30(11):1331-4. doi: 10.1097/01.brs.0000164099.92112.29. PMID 15928561
- [Background] Ferreira-Valente MA, Pais-Ribeiro JL, Jensen MP. Validity of four pain intensity rating scales. Pain. 2011 Oct;152(10):2399-2404. doi: 10.1016/j.pain.2011.07.005. PMID 21856077
- [Background] Ostelo RW, Deyo RA, Stratford P, Waddell G, Croft P, Von Korff M, Bouter LM, de Vet HC. Interpreting change scores for pain and functional status in low back pain: towards international consensus regarding minimal important change. Spine (Phila Pa 1976). 2008 Jan 1;33(1):90-4. doi: 10.1097/BRS.0b013e31815e3a10. PMID 18165753
- [Background] Waterschoot FPC, Dijkstra PU, Hollak N, de Vries HJ, Geertzen JHB, Reneman MF. Dose or content? Effectiveness of pain rehabilitation programs for patients with chronic low back pain: a systematic review. Pain. 2014 Jan;155(1):179-189. doi: 10.1016/j.pain.2013.10.006. Epub 2013 Oct 14. PMID 24135435
- [Background] Navani A, Manchikanti L, Albers SL, Latchaw RE, Sanapati J, Kaye AD, Atluri S, Jordan S, Gupta A, Cedeno D, Vallejo A, Fellows B, Knezevic NN, Pappolla M, Diwan S, Trescot AM, Soin A, Kaye AM, Aydin SM, Calodney AK, Candido KD, Bakshi S, Benyamin RM, Vallejo R, Watanabe A, Beall D, Stitik TP, Foye PM, Helander EM, Hirsch JA. Responsible, Safe, and Effective Use of Biologics in the Management of Low Back Pain: American Society of Interventional Pain Physicians (ASIPP) Guidelines. Pain Physician. 2019 Jan;22(1S):S1-S74. PMID 30717500
- [Background] Pettine KA, Suzuki RK, Sand TT, Murphy MB. Autologous bone marrow concentrate intradiscal injection for the treatment of degenerative disc disease with three-year follow-up. Int Orthop. 2017 Oct;41(10):2097-2103. doi: 10.1007/s00264-017-3560-9. Epub 2017 Jul 26. PMID 28748380